CLINICAL TRIAL: NCT02346539
Title: Effect of Nicotine on Brain Reward Pathways
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mclean Hospital (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Amy C. Janes, Assistant Professor/Neuroscientist, Mclean Hospital
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 2014P002495-01; 5K01DA029645-04 (NIH)
Record Dates: First submitted 2015-01-14; First posted 2015-01-27 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-03

CONDITIONS: Depressive Disorder
Keywords: Nicotine; Depression
MeSH Terms: conditions — Depressive Disorder; Depression | interventions — Tobacco Use Cessation Devices

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nicotine (Experimental): 2mg of nicotine in the form of a nicotine polacrilex lozenge will be administered orally, one time.
  4mg of nicotine in the form of a nicotine polacrilex lozenge will be administered orally, one time.
  Interventions: Drug: Nicotine polacrilex
- Placebo (Placebo Comparator): Placebo comparator
  Interventions: Drug: Nicotine polacrilex

INTERVENTIONS:
Drug: Nicotine polacrilex — Single Acute dose
  Other Names: Nicotine lozenge

SUMMARY:
The investigators will determine whether an acute dose of nicotine, in the form of the nicotine lozenge, impacts brain and behavioral measures of mood and reward responsiveness in individuals with major depressive disorder.

ELIGIBILITY:
Inclusion Criteria for subjects with Major Depressive Disorder:

1. Provide written informed consent;
2. Both genders and all ethnic origins, age between 18 and 45;
3. Meet DSM-IV diagnostic criteria for MDD (diagnosed with the use of the SCID);
4. A baseline HAM-D score of 16 or greater;
5. Absence of pregnancy;
6. Absence of any psychotropic medication for at least 2 weeks:

   1. 6 weeks for fluoxetine
   2. 6 months for neuroleptics
   3. 2 weeks for benzodiazepines
   4. 2 weeks for any other antidepressants

Inclusion Criteria for Healthy Controls

1. Absence of medical, neurological, and psychiatric illness (including alcohol and substance abuse); as assessed by subject history and a structured clinical interview (SCID);
2. Provide written informed consent;
3. Both genders and all ethnic origins, age between 18 and 45;
4. Absence of any medications for at least 3 weeks;
5. Absence of pregnancy.

Exclusion Criteria:

1. Subjects with suicidal ideation where outpatient treatment is determined unsafe. These patients will be immediately referred to a licensed psychologist or psychiatrist to determine the appropriate clinical treatment;
2. Serious or unstable medical illness
3. Lifetime history of seizure disorder;
4. Lifetime history or current diagnosis of any of the following DSM-IV psychiatric illnesses: organic mental disorder, schizophrenia, schizoaffective disorder, delusional disorder, psychotic disorders not otherwise specified, bipolar disorder, ADHD, patients with mood congruent or mood incongruent psychotic features; simple phobia, social anxiety disorder and generalized anxiety disorders will be allowed only if secondary to MDD;
5. Patients with a lifetime history of electroconvulsive therapy (ECT);
6. Failure to meet standard MRI safety requirements;
7. May not have used any nicotine product in the past year; must report fewer than 20 lifetime uses of nicotine
8. Must have an expired carbon monoxide level of less than or equal to 10 ppm.
9. Use of anticholinergic drugs in the past week
10. Any past or present history of cardiac problems including known arrhythmias, acute coronary syndrome, or ischemic heart disease
11. Uncontrolled hypertension
12. History of substance abuse in the past 6 months (other than caffeine), self-reported use of marijuana in past month, or history of treatment with methadone
13. Heavy caffeine users (consume greater than 500 mg on a regular or daily basis)
14. Subjects that cannot speak English

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2015-02; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
Change from Placebo in functional magnetic resonance imaging (fMRI) BOLD Response | Participants will be assessed during 2 fMRI scanning sessions, an expected average of 2 weeks.
  Nicotine will enhance the fMRI BOLD response to monetary reinforcers relative to placebo administration

CONTACTS AND LOCATIONS:
Overall Officials: Amy Janes, Ph.D, Principal Investigator — Mclean Hospital
Locations (1):
- McLean Hospital, Belmont, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang KS, Brown K, Frederick BB, Moran LV, Olson D, Pizzagalli DA, Kaiser RH, Janes AC. Nicotine acutely alters temporal properties of resting brain states. Drug Alcohol Depend. 2021 Sep 1;226:108846. doi: 10.1016/j.drugalcdep.2021.108846. Epub 2021 Jun 24. PMID 34198131